CLINICAL TRIAL: NCT06825871
Title: Automated Inhaler Monitoring for Asthma Medication Usage
Acronym: AIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Respiratory Analytics Ltd (Unknown)
Responsible Party: Principal Investigator, Wanda Phipatanakul, S. Jean Emans, MD, Professor of Pediatrics at Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00049452
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Asthma; Inhalers; Quality Control; Digital Health
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention group (Experimental): Participants will use the aflo™ digital platform, which includes an electronic inhaler sensor, a mobile application, and a clinician portal. The platform provides real-time feedback on inhaler technique and sends medication reminders to improve adherence. Participants will also receive daily symptom tracking prompts and monthly Asthma Control Test (ACT) assessments.
  During the study, participants will:
  * Attach the aflo™ sensor to their metered-dose inhaler (MDI) and use it with or without a spacer, based on their prescribed regimen.
  * Complete at least one supervised inhalation session during the baseline visit to ensure proper use of the sensor.
  * Use the aflo™ mobile app to log asthma symptoms, medication usage, and track reminders.
  * Participate in two clinic visits (at baseline and study completion) and two follow-up phone calls (at weeks 4 and 8) to monitor progress.
  Interventions: Device: Smart Inhaler Monitoring Platform for Asthma Management

INTERVENTIONS:
Device: Smart Inhaler Monitoring Platform for Asthma Management — The intervention utilizes the aflo™ digital platform, a comprehensive system designed to improve asthma management through advanced technology. It integrates the following components:
  1. Electronic Inhaler Sensor: The sensor attaches to a metered-dose inhaler (MDI) and a spacer (if applicable) to automate and provide feedback on the six critical steps of proper inhaler technique, such as shaking the inhaler, breathing out, inhaling slowly, and holding the breath. The sensor also records and stores medication usage data securely.
  2. Mobile Application: The app delivers real-time notifications and feedback on inhaler technique, sends reminders for daily controller medication, tracks asthma symptoms, and provides monthly Asthma Control Test (ACT) assessments. It also offers reminders for spacer cleaning and customizable alerts for caregivers.
  3. Clinician Portal: Data collected from the sensor and app is accessible via a secure clinician portal, enabling healthcare providers to monitor pa

SUMMARY:
The goal of this clinical trial is to evaluate the aflo™ digital platform's ability to improve inhaler use technique and asthma control for children, adolescents, and adults with uncontrolled asthma. The main questions the trial aims to answer are:

1. Does the platform improve medication adherence and inhaler technique, as measured by the Inhaler Proficiency Score (IPS)?
2. Does the aflo™ platform improve asthma control, as measured by changes in the Asthma Control Test (ACT) and lung function tests (FEV1, PEF)?

Participants will:

* Use the aflo™ sensor with their asthma inhaler to receive real-time feedback on technique and medication adherence reminders.
* Track asthma symptoms and quality of life through a mobile app.
* Complete assessment visits and surveys at the start and end of the 3-month study and 2 interim asthma assessment phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. Youth or adult with a diagnosis of persistent asthma by a physician.
2. Evidence of uncontrolled asthma as defined by an FEV1/FVC ratio of less than 80% by an asthma provider within the past 3 months, all while on controller asthma therapy.
3. Females or males between the ages of 10 years and older
4. Participant or caregiver must have an Apple and/or Android smart phone with operating system 4.3 or above and data plan for the duration of the study period

Exclusion Criteria:

1. Participants with other cardiac, pulmonary with exception of asthma, neuromuscular disorders that impact breathing, or other conditions that hinder patient to perform spirometry.
2. Participants with severe neurobehavioral, neurodevelopmental, or psychiatric disorders requiring special assistance
3. The participant's guardian or the patient has comprehension or language difficulties that prevent understanding of study materials (available in English) or effective training on the app or device.
4. Patients are currently receiving biologic therapies for asthma management or other allergic diseases.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the participants' Inhaler Proficiency Score (IPS) Following Aflo™ Platform Usage at 3 Month | From enrollment to the end of intervention period at 12 weeks
  Inhaler Proficiency Score (IPS) is a validated, composite score that assesses the accuracy and consistency of inhaler technique, including steps such as inhaler preparation, actuation timing, inhalation depth, and breath hold. Scores range from 0 to 10, with higher scores indicating greater inhaler technique proficiency. Scores will be recorded at baseline and again after 3 months of using the Aflo™ digital platform, which provides step-by-step guidance and real-time feedback on inhaler technique. The outcome measure reflects the mean change in IPS from baseline to the 3-month follow-up to evaluate the effectiveness of the intervention.

SECONDARY OUTCOMES:
Evaluation of the aflo™ Platform for Improving Asthma Control Using ACT Scores | From enrollment to the end of intervention period at 12 weeks
  This study assesses the impact of the aflo™ platform on asthma control, measured by changes in Asthma Control Test (ACT) scores. The ACT is a validated questionnaire used to evaluate asthma management, with scores ranging from 5 (poor control) to 25 (complete control). Participants will use the aflo™ platform, which provides real-time inhaler usage feedback via a connected device and mobile app. ACT scores will be collected at baseline and after the intervention to determine the platform's effectiveness in improving asthma outcomes.
Impact of the aflo™ Platform on Health-Related Quality of Life and Clinical Outcomes in Asthma | From enrollment to the end of intervention period at 12 weeks
  This study evaluates secondary outcomes of the aflo™ platform, including maximal percent changes in self- and parent-reported health-related quality of life using the St. George's Respiratory Questionnaire (SGRQ). Additional clinical outcome measures, such as lung function and symptom changes, will also be assessed. These measures aim to further understand the platform's effect on asthma management beyond asthma control.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No